CLINICAL TRIAL: NCT00201539
Title: Double Bedtime Dosing During Immediate-release Morphine Administration to Cancer Patients: A Randomized, Double-blind Cross-over Comparison of a Double Bedtime Dose Ver-sus Two Standard Doses at Bedtime and at Night
Brief Title: Double Bedtime Dosing During Immediate-release Morphine Administration to Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OPI 02/001
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: analgesics, opioid/pharmacokinetics; humans; morphine/therapeutic use*; neoplasms; pain/drugtherapy
MeSH Terms: conditions — Neoplasms | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- double dose once (Active Comparator): double dose immediate-release oral morphine at bedtime in cancer patients, placebo after 4 hours
  Interventions: Drug: double dose Morphine; Drug: placebo
- single dose twice (Experimental): single dose immediate-release oral morphine at bedtime in cancer patients, second single dose after 4 hrs
  Interventions: Drug: single dose Morphine

INTERVENTIONS:
Drug: single dose Morphine
  Arms: single dose twice
Drug: double dose Morphine
  Arms: double dose once
Drug: placebo — purchased from the manufacturer of morphine tablets (Nycomed Pharma, Oslo, Norway)
  Arms: double dose once

SUMMARY:
This is a double -blind randomized crossover study to provide evidence for the expert advice based recommendation of the Expert Working Group of the European Association for Palliative Care (EAPC) that patients during treatment with IR morphine are given a double dose at bed-time that replaces the next 4-hourly dose during night. In addition to the primary, blinded clinical part of the study, an experimental part is also included. This part consists of two open study days were morphine IR is given in the same fashion as the clinical study. The aim is to study whether pharmacokinetic data supports the clinical data.

The use of a double-bedtime IR morphine dose is equal to regularly scheduled IR morphine every 4-hour during night in respect to pain relief during night for patients with pain caused by malignant disease

DETAILED DESCRIPTION:
PROTOCOL

Double bedtime dosing during immediate-release morphine administration to cancer patients:

A randomized, double-blind cross-over comparison of a double bedtime dose versus two standard doses at bedtime and at night

Introduction

Oral morphine is recommended by the World Health Organization for pain control in moderate or strong cancer pain 1. At our hospital we use the practice recommended by the Expert Working Group of the European Association for Palliative Care for introduction of strong opioids with titration with immediate-release (IR) morphine dosed every 4 hour until an optimal balance between analgesia and side effects is achieved. After the optimal daily dose is defined slow-release (SR) morphine in the same total daily morphine dose is started 2. One of the features of the EPAC guidelines is that patients during treatment with IR morphine are given a double bed-time that replaces the next 4-hourly dose during night 2. The rationale behind this recommendation is that giving a double dose will prolong duration of morphine analgesia and eliminate the need for awaking the patient during night. However, this recommendation is based on expert opinion and not evidence from clinical studies 2. Todd et al. has recently presented results that challenge this approach from a cross-over study in which the patients received either a double bedtime dose or regular doses every 4-hour 3. This study showed that patients receiving a double bedtime dose reported more pain, more use of rescue medications and reported inferior sleep quality compared to patients receiving regularly scheduled doses. A limitation of this study was that they did not perform the study blinded and thus consequently the results are subject to bias. It is a need for a placebo-controlled study before the evidence carries enough weight to change current recommendations.

Besides a clinical study it is also relevant to obtain pharmacokinetic observations during double bedtime and regularly IR morphine dosing. Repeated blood sampling will disturb the patients during night and hence confound the clinical observations (e.g. sleep quality). Consequently, the blood samples will not be obtained in the same dosing interval where the clinical data are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant disease
* Age more than 18 year
* Regular use of oral morphine or pain that indicates start of opioids for moderate or severe pain according to the WHO guidelines for treatment of cancer pain

Exclusion criteria

* Known morphine intolerance
* History of drug abuse
* Decreased gastrointestinal uptake of oral medications
* Pregnancy or breast-feeding
* General health condition, psychiatric disease or cognitive function failure giving that the patient is not competent to complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-04; Primary Completion 2006-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variable
Patient rating of average pain intensity during night measured on a 11-point nu-meric rate scale

SECONDARY OUTCOMES:
Secondary efficacy variables
Pain rating of "pain now" before scheduled morning dose measured on a 11-point numeric rate scale
Number of rescue opioid medications during night
Patient overall rating of sleep quality during night measured on a 11-point nu-meric rate scale
Number of episodes being awake during night
Rating of pain intensity measured on a 11-point numeric rate scale when being awake at night
Overall rating of side effects (nausea, xerostomia, tiredeness) during night meas-ured on 11-point numeric rate scales
Pain preference of treatments:
Time-course of serum concentrations of morphine, morphine-6-glucurnide (M6G) and morphine-3-glucuronide (M3G) will be obtained during two 4-hourly dose intervals and one 8-hour dose interval after a double dose administration
Pharmacodynamic time-course efficacy of opioids measured by pupillometri will be obtained during two 4-hourly dose intervals and one 8-hour dose interval after a double dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Paal Klepstad, Md,PhD, Principal Investigator — St.Olavs University Hospital, Norway
Locations (2):
- Norway (2):
  - The Norwegian Univeristy of tecknology and science, Trondheim, Trondheim
  - St Olavs University Hospital, Trondheim

REFERENCES:
- [Result] Dale O, Piribauer M, Kaasa S, Moksnes K, Knobel H, Klepstad P. A double-blind, randomized, crossover comparison between single-dose and double-dose immediate-release oral morphine at bedtime in cancer patients. J Pain Symptom Manage. 2009 Jan;37(1):68-76. doi: 10.1016/j.jpainsymman.2007.12.016. Epub 2008 May 27. PMID 18504090